CLINICAL TRIAL: NCT07058571
Title: Lifestyle Intervention for Veterans With Blood Cancer: Tele-Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1823598
Record Dates: First submitted 2025-05-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Blood Cancers
Keywords: Physical Activity; Exercise; Tele-oncology; Blood Cancer
MeSH Terms: conditions — Hematologic Neoplasms; Motor Activity | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): All veterans in the intervention group (e.g., total N) will engage in 12 week telehealth mediated exercise intervention. Veterans will also have the opportunity to undergo a centralized dietary consultation and recommendations (by a Leukemia and Lymphoma Society (LLS) member).
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION

INTERVENTIONS:
Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — Participating Veterans will engage in bi-weekly, telehealth mediated resistance exercise session. Aerobic exercise will be monitored passively through FitBit data collection. Telehealth exercise sessions will last approximately 45-90 minutes pending the individual Veteran's progress. Participants will also undergo a one-time dietary consultation and recommendations by a Leukemia and Lymphoma Society (LLS) member.

SUMMARY:
Background. This study aims to evaluate the effectiveness of a telehealth-mediated lifestyle intervention program tailored for veterans with blood cancer, focusing on improving health-related quality of life, mental health, and pain outcomes. The hypothesis posits that the telehealth-delivered program will lead to significant improvements in these areas, specifically targeting veterans undergoing treatment or in post-treatment phases.

Objective. Recognizing the unique experiences of veterans, especially those in rural or underserved regions, this study seeks to provide insights into the feasibility and impact of telehealth-based lifestyle interventions for this distinct population.

Methods. The pilot trial will enroll 30 veterans from the H. John Heinz III VA. Participants will complete baseline web-based surveys assessing demographics, occupational performance, and telehealth preparedness. The intervention comprises progressive resistance and aerobic exercises delivered via telehealth by a health coach, starting with a live supervised session followed by regular remote sessions. Each participant will engage in exercise sessions coordinated through the Veteran's Video Connect (VVC) application, with ongoing communication facilitated via email. This setup allows the health coach to adjust exercise intensity based on real-time symptom feedback.

To address potential technology literacy biases, the VVCMatch assessment will categorize veterans as "technology prepared" or in need of additional education. Those requiring support will receive guidance on using the VVC app before starting the intervention. Additionally, participants will receive dietary consultations from the Leukemia and Lymphoma Society, independent of the research team.

Outcome measures include assessments of symptoms, fatigue, function, mental health, and pain, along with evaluations of the intervention's usability through surveys on perceived usefulness and ease of use. These assessments aim to detect meaningful changes and ensure the intervention's effectiveness and acceptability among veterans.

DETAILED DESCRIPTION:
Background. Since the changes in care delivery brought about by the COVID-19 pandemic, around 12% of outpatient cancer care visits are now conducted via telehealth. This approach, known as tele-oncology, offers cancer patients more efficient, convenient, and crucially, accessible care options. For VA populations, tele-oncology provides opportunities for follow-up post-diagnosis visits, visits while undergoing therapy (replacing in-person visits on chemotherapy days), and ongoing health surveillance. Variations in digital literacy among veterans can introduce bias in essential research on telehealth-delivered care interventions. To tackle this issue, our team has created and tested the VVCMatch, a tailored telehealth readiness tool. The VVCMatch is intended to proactively identify various barriers to tele-oncology that veterans may face, such as communication impairments and cognitive changes related to chemotherapy or hormonal therapy, including memory, mental flexibility, and processing challenges.

The proposed study aims to assess the efficacy of a telehealth-mediated lifestyle intervention program specifically designed for veterans with blood cancer. The primary focus is on evaluating improvements in health-related quality of life, mental health, and pain outcomes. This initiative acknowledges the unique experiences and challenges faced by veterans, who constitute a distinct population with specific needs, particularly those residing in rural or underserved areas. We hypothesize that the telehealth-delivered lifestyle intervention will result in significant enhancements in health-related quality of life, reduction in depressive symptoms, improved functional capacity, and decreased pain levels among the veteran participants. Such improvements are crucial for this demographic, as they often face barriers to accessing consistent, high-quality healthcare services.

Methods. This pilot trial will enroll 30 veterans from the H. John Heinz III VA, including those currently receiving treatment (such as chemotherapy or radiation therapy) and those in post-treatment stages. This inclusive approach is intended to increase recruitment feasibility and provide comprehensive insights across different treatment timelines. Baseline measurements will be collected through web-based surveys that evaluate demographics, occupational performance via the Canadian Occupational Performance Measure, and telehealth preparedness using the VVCMatch assessment.

The intervention itself is composed of two main components: progressive resistance and aerobic exercises. These will be delivered through a distance model facilitated by a health coach. The intervention begins with an initial supervised live exercise session conducted via telehealth, followed by regular remote sessions lasting 30 to 45 minutes each. These sessions are carried out via telehealth through the Veteran's Video Connect (VVC) application, with scheduling tailored to each participant's availability. Between sessions, communication is maintained through email, allowing for the exchange of information regarding session schedules and graphical progress reports.

A critical feature of this study is its adaptability to the participants' real-time needs. The health coach can modify exercise intensity based on daily symptom assessments, ensuring that each session is both effective and safe. This responsiveness is particularly important given the fluctuating nature of symptoms in individuals with blood cancer. To address potential disparities in technology literacy, the VVCMatch assessment will categorize participants into either a "technology prepared" or "technology education" group. Those identified as needing additional support will receive comprehensive telehealth education, including a walkthrough of the VVC application, to ensure they can fully engage with the intervention.

In addition to the physical activity component of exercise, participants will also have access to dietary consultations provided by the Leukemia and Lymphoma Society (LLS). This service underscores the holistic approach of the intervention, addressing both physical and dietary aspects of health.

Outcome measures include a range of assessments conducted at baseline and post-intervention. These encompass symptoms (using the VA Symptom Assessment Scale), fatigue (measured by the Global Fatigue Index), functional capacity (assessed via the PROMIS-Physical Function Cancer Item Bank), mental health (evaluated with the Four-Item Patient Health Questionnaire for Anxiety and Depression), and pain (measured using the Numeric Pain Rating Scale and the McGill Pain Questionnaire Short-Form). The intervention's usability will also be assessed using the Technology Acceptance Model, focusing on perceived usability, usefulness, and ease of use.

Overall, this study aims to provide valuable insights into the feasibility and impact of telehealth-based lifestyle interventions for veterans with blood cancer, potentially offering a scalable model to enhance the quality of life for this underserved population.

ELIGIBILITY:
Inclusion Criteria:

* Living with blood cancer
* Physically willing and able to perform 30-90 minutes of exercise a minimum of 2 times per week

Exclusion Criteria:

* Veterans who are unable to perform 30-90 minutes of exercise twice a week
* Veterans with significant disabilities related to balance or motion that would cause a safety risk
* Veterans without a smart personal device (smart phone, tablet, or computer) and internet connection (for example, cellular or WIFI connection)
* Veterans who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04-03 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
VVCMatch telehealth preparedness measure (5 Minute Montreal Cognitive Assessment component) | Baseline
  The Veteran's Video Connect (VVC)Match assesses Veteran's telehealth preparedness by considering their cognitive, physical, and digital literacy ability levels. The VVCMatch incorporates the 5-minute telephone Montreal Cognitive Assessment, followed by 28 self-report items.
Demographics Form | Baseline
Global Fatigue Index | Baseline and 12 weeks follow-up
  A 15 item self-report assessment to gauge the impact that fatigue has has on and individual's day-to-day life.
The Numeric Pain Rating Scale Instructions | Baseline and 12 weeks follow-up
  An assessment that investigates the severity of an individual's current level of pain, and the lowest and highest level of pain they experienced in the past 24 hours.
Four-Item Patient Health Questionnaire for Anxiety and Depression | Baseline and 12 weeks follow-up
  A 4-item, self-report measure assessing the frequency of mental health symptoms across a 2-week period.
Numeric Pain Rating Scale and McGill Pain Questionnaire Short-Form | Baseline and 12 weeks follow-up
  A 15 item, self-report measure asking about the location and type of an individuals current pain level.
PROMIS-Physical Function Cancer Item Bank | Baseline and 12 weeks follow-up
  A 45 item, self-report measure of physical function, with responses ranging from 1 (Unable to do) to 5 (Without any difficulty).

SECONDARY OUTCOMES:
Technology Acceptance Model surveys | 12 weeks follow-up (Post-Intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mounier NM, Abdel-Maged AE, Wahdan SA, Gad AM, Azab SS. Chemotherapy-induced cognitive impairment (CICI): An overview of etiology and pathogenesis. Life Sci. 2020 Oct 1;258:118071. doi: 10.1016/j.lfs.2020.118071. Epub 2020 Jul 14. PMID 32673664
- [Background] Jiang CY, El-Kouri NT, Elliot D, Shields J, Caram MEV, Frankel TL, Ramnath N, Passero VA. Telehealth for Cancer Care in Veterans: Opportunities and Challenges Revealed by COVID. JCO Oncol Pract. 2021 Jan;17(1):22-29. doi: 10.1200/OP.20.00520. Epub 2020 Sep 24. PMID 32970512
- [Background] Rapid Growth in Telehealth for Cancer Care - NCI. Published March 9, 2022. Accessed May 31, 2023. https://www.cancer.gov/news-events/cancer-currents-blog/2022/pandemic-telehealth-surge-cancer-care